CLINICAL TRIAL: NCT04413253
Title: Intracanalicular Dexamethasone Used in Conjunction With Xiidra (Lifitegrast Ophthalmic Solution) for the Treatment of Signs and Symptoms of Dry Eye Disease as Compared to Xiidra Alone
Brief Title: Xiidra vs. Xiidra + Dextenza Treatment for Dry Eye Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: Eye Surgeons of Indiana (Network)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: The DAMON Study
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast; Ophthalmic Solutions; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xiidra Only Group (Active Comparator): Patients with dry eye disease Xiidra only
  Interventions: Drug: Lifitegrast 5% Ophthalmic Solution
- Xiidra + Dextenza Group (Experimental): Patients with dry eye disease Xiidra + Dextenza
  Interventions: Drug: Dexamethasone Intracanalicular Insert, 0.4mg with Lifitegrast 5% Ophthalmic Solution

INTERVENTIONS:
Drug: Lifitegrast 5% Ophthalmic Solution — To reduce signs and symptoms of dry eye disease
  Other Names: Xiidra
  Arms: Xiidra Only Group
Drug: Dexamethasone Intracanalicular Insert, 0.4mg with Lifitegrast 5% Ophthalmic Solution — To determine the outcomes of reduction of signs and symptoms of dry eye disease with DEXTENZA as an added therapy, in addition to Xiidra therapy.
  Other Names: Dextenza; Xiidra
  Arms: Xiidra + Dextenza Group

SUMMARY:
To evaluate the benefit of treatment with a physician administered intracanalicular dexamethasone insert in patients with dry eye who are beginning treatment with Xiidra (lifitegrast ophthalmic solution) to reduce the signs and symptoms of dry eye disease.

DETAILED DESCRIPTION:
This prospective study will use a fellow-eye design for 20 participants, 40 eyes. All eyes will receive bilateral Xiidra. The most symptomatic eye will be selected to receive DEXTENZA® insertion on the day Xiidra is prescribed (study eye), while the other eye will be assigned to receive sham punctum dilation (control eye). If there is no obvious symptomatic difference, the right eye will receive the intracanalicular insert. The study group will consist of 20 eyes receiving DEXTENZA® insertion. The control group will consist of 20 eyes receiving sham punctum dilation. Thus, for every eye in the study group, there will be a paired eye with similar baseline characteristics in the control group sourced from the same participant. This fellow-eye design allows for greater control of potential confounders tied to participants' systemic and ocular health.

ELIGIBILITY:
Inclusion Criteria:

A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

* 18 years of age or older
* Signs and symptoms of DED
* Consent to treat with topical immunomodulator
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

* Patients under the age of 18.
* Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Altered nasolacrimal flow of either acquired, induced, or congenital origin
* Hypersensitivity to dexamethasone
* Patients who have been on topical immunomodulating agents in the previous 3 months to their baseline visit
* Patient being treated with either topical, oral, or intravenous immunosuppressive agents, immunomodulating agents, or steroid (including NSAIDS)
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Mean change in ocular surface staining | Assessed at Baseline, Week 1, Week 2, Week 4 and Week 12 Visit
  As measured by sodium fluorescein and lissamine green
Patient Preference for therapy | Assessed at Week 12 Visit
  As measured by COMTOL Survey

SECONDARY OUTCOMES:
Mean change in MMP-9 | Assessed at Baseline, Week 1, Week 2, Week 4 and Week 12 Visit
  As measure by InflammaDry
Mean change in tear break-up time (TBUT) | Assessed at Baseline, Week 1, Week 2, Week 4 and Week 12 Visit
  As measured by TBUT testing
Mean change in conjunctival injection | Assessed at Baseline, Week 1, Week 2, Week 4 and Week 12 Visit
  As measured on a scale of 0-4 and graded by the physician
Change from baseline in meibomian gland scores (expressibility and quality) | Assessed at Baseline, Week 1, Week 2, Week 4 and Week 12 Visit
  As measured on a grading scale 1 to 4 and graded by the physician
Mean change in tear osmolarity | Assessed at Baseline, Week 1, Week 2, Week 4 and Week 12 Visit
  As measured by Tear Lab
Mean change in DEQ-5 | Assessed at Baseline, Week 1, Week 2, Week 4 and Week 12 Visit
  As measured by the DEQ-5 Questionnaire
Mean change in Best-corrected Visual Acuity (BCVA) | Assessed at Baseline, Week 1, Week 2, Week 4 and Week 12 Visit
  As measure by ETDRS

CONTACTS AND LOCATIONS:
Overall Officials: Damon Dierker, OD, FAAO, Principal Investigator — Eye Surgeons of Indiana
Locations (1):
- Eye Surgeons of Indiana, Indianapolis, Indiana, United States